CLINICAL TRIAL: NCT06231888
Title: Difference Between Pressing and Vacuum Techniques in Fabrication of Orthodontic Aligners in Cases With Crowding: A Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abd El-Ghafour, Lecturer, Department of Orthodontics, Cairo University
Other Study IDs: 005
Record Dates: First submitted 2024-01-13; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Orthodontic Aligners
MeSH Terms: interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Press
  Interventions: Device: Aligner
- Vacuum
  Interventions: Device: Aligner

INTERVENTIONS:
Device: Aligner — Orthodontic alginer

SUMMARY:
This cross sectional study is aiming to compare 2 methods of clear aligner fabrication.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary arch with crowding.
* Full permanent dentition.

Exclusion Criteria:

* Missing teeth.
* Dental restorations.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Maxillary arch with moderate crowding.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Maxillary arch dimensions | 6 months
  Arch lengths, Arch widths and each tooth size will be measured and compared between the 2 groups.

SECONDARY OUTCOMES:
Model superimposition | 6 months
  Superimposition of the models from the 2 groups will be done and then map difference will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided